CLINICAL TRIAL: NCT03696173
Title: Comparative Safety of Biologic Disease-modifying Treatment Initiation With Abatacept in Rheumatoid Arthritis: A Real-world Population-based Observational Study
Brief Title: Safety Study of Abatacept in Rheumatoid Arthritis Participants
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM101-605
Record Dates: First submitted 2018-10-03; First posted 2018-10-04 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2018-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants taking abatacept
  Interventions: Other: Non-Interventional
- Participants taking abatacept with methotrexate
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — Non-Interventional
  Groups: Participants taking abatacept
Other: Non-Interventional — Non-Interventional
  Groups: Participants taking abatacept with methotrexate

SUMMARY:
A observational study to assess whether biologic disease-modifying (BDM) treatment initiation with abatacept for rheumatoid arthritis is associated with an increased risk of serious infection and cancer

ELIGIBILITY:
Inclusion Criteria:

* Patient initiates BDM treatment with at least one claim for the treatment. Patients will be presumed to be new users of a treatment if there is no claim for the drug or any other BDM in the 180 days prior to the cohort entry date
* Patient has at least two diagnoses for RA in the patient's history prior to and including the entry date or within the 180 days after the entry date
* Patient is aged 18 years or older on the entry date
* Patient was enrolled in the database for at least 180 days before the entry date

Exclusion Criteria:

* Patient is younger than 18 years on the entry date
* Patients who receive abatacept and another biologic simultaneously
* Patients who have an outcome diagnosis in the baseline period will be excluded from the cohort analyses for that outcome

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rheumatoid arthritis (RA) participant, population-based cohort study approach within the US-based Truven MarketScan population and Supplemental US Medicare database
Sampling Method: Probability Sample
Enrollment: 5800 (Estimated)
Dates: Start 2015-12-17 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2018-06-29 (Actual)

PRIMARY OUTCOMES:
Incidence of increased risk of serious infection while taking abatacept | Approximately 7 years
  With methotrexate
Incidence of malignancy while taking abatacept | Approximately 7 years
  With methotrexate
Incidence of increased risk of serious infection while taking abatacept | Approximately 7 years
  Without methotrexate
Incidence of malignancy while taking abatacept | Approximately 7 years
  Without methotrexate

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Princeton, New Jersey, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx